CLINICAL TRIAL: NCT03352804
Title: Are the Patients Having Pets at Greater Risk of Carrying Multidrug Resistance Bacteriae?
Acronym: BRANITRANS
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO17041*
Record Dates: First submitted 2017-11-17; First posted 2017-11-24 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Multidrug Resistance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients hospitalized in internal medicine ward: Patients included are patients hospitalized in internal medicine ward.
  Interventions: Other: Screening of MDR Bacteriae

INTERVENTIONS:
Other: Screening of MDR Bacteriae — questionnaire will be filled by every patient

SUMMARY:
Introduction : The multidrug resistance (MDR) Bacteriae are growing and are a public health problem. The known risk factors to be expanding of MDR Bacteriae are: taken antibiotics, hospitalization, journey in a country at risk. Other risk factors are emitted in hypothesis as the presence of pets.

Aim : The primary objective is to study the association between the presence of a pet and the presence of a MDR bacteria. Methods : Cross sectional study will be performed in Reims University hospital in internal medicine ward.

DETAILED DESCRIPTION:
Introduction : The multidrug resistance (MDR) Bacteriae are growing and are a public health problem. The known risk factors to be expanding of MDR Bacteriae are: taken antibiotics, hospitalization, journey in a country at risk. Other risk factors are emitted in hypothesis as the presence of pets.

Aim : The primary objective is to study the association between the presence of a pet and the presence of a MDR bacteria.

Methods : Cross sectional study will be performed in Reims University hospital in internal medicine ward. Within the framework of the management of patients in internal medicine ward, all the hospitalized patients have systematically a screening of MDR Bacteriae. A questionnaire will be put handed to all the patients during their hospitalization as soon as they will be able to answer it. They will be informed about the objectives of the study. If the patient agrees to participate in the study, the questionnaire will be filled by every patient. It includes essentially closed questions and some open questions. A descriptive analysis will be performed. Bivariate analysis will be performed to investigate the relation between the presence of a pet and the presence of a MDR bacteria and clinical variables Multivariate logistic regression will be performed to investigate the factors independently related to the presence of a MDR bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were screened for MDR bacteria
* Patients who accepted to participate in the study
* >18yo

exclusion criteria :

* Patient hospitalized before admission in our ward and having acquired a MDR bacteria in the course of care.
* Patients coming from nursing home or institutionalized patients
* Patient who cannot communicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in internal medicine ward of Reims University hospital
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Association between the presence of a pet and the presence of a MDR bacteria | Day0

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided